CLINICAL TRIAL: NCT02941185
Title: Multi-dose Vitamin D Supplementation in Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Ozlem Bozkurt, MD, Neonatology fellow, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZTB2015
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Vitamin D Deficiency; Preterm Infants
MeSH Terms: conditions — Vitamin D Deficiency

ARMS (3):
- Devit-3 Oral Drop 400 IU (Other): supplemented with oral Vitamin D 400 IU/day (Devit-3 Oral Drop, 50000 IU/15 ml, Deva Company, Turkey) started when achieved 75%of total nutrition by enteral feedings and continued until 36 weeks postmenstrual age
  Interventions: Drug: Devit-3 Oral Drop
- Devit-3 Oral Drop 800 IU (Active Comparator): Devit-3 Oral Drop 800 IU once daily by oral route started when achieved 75%of total nutrition by enteral feedings and continued until 36 weeks postmenstrual age
  Interventions: Drug: Devit-3 Oral Drop
- Devit-3 Oral Drop 1000 IU (Active Comparator): Devit-3 Oral Drop1000 IU once daily by oral route started when achieved 75%of total nutrition by enteral feedings and continued until 36 weeks postmenstrual age
  Interventions: Drug: Devit-3 Oral Drop

INTERVENTIONS:
Drug: Devit-3 Oral Drop

SUMMARY:
Preterm newborns are born with lower vitamin D stores. Although vitamin D supplementation is recommended there is no consensus regarding the adequate dose of supplementation for preterm infants.

DETAILED DESCRIPTION:
Vitamin D is a fat-soluble vitamin that is either taken by dietary sources or synthesized upon exposure to sun light. Although major function is on bone metabolism, in recent years other effects of Vitamin D attracted attention. Low neonatal vitamin D levels were reported to be associated with increased risk of respiratory distress syndrome (RDS), bronchopulmonary dysplasia (BPD) and sepsis.

Vitamin D level in the fetus and the newborn is mostly dependent on maternal vitamin D levels. Most of the vitamin D is transferred to the fetus during third trimester and as a result preterm newborns especially those with <32 weeks gestational age are born with lower vitamin D stores. But there is no consensus regarding the adequate dose of vitamin D supplementation for preterm infants. The American Academy of Pediatrics recommends supplementation of 200-400 IU/d vitamin D for preterm infants. And the European Society of Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) recommends 800-1000 IU/d vitamin D supplementation for preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age 24 to 32 weeks who achieved at least 75% of total nutrition by enteral feedings in postnatal 2 weeks

Exclusion Criteria:

* perinatal asphyxia,
* major congenital or chromosomal anomalies,
* those with no expectation of survival in first 2 weeks
* those that total parenteral nutrition was not ceased by the first 2 weeks

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Serum concentration of 25(OH) D at 36 weeks postmenstrual age. | 36 weeks
Prevalence of vitamin D deficiency at 36 weeks postmenstrual age. | 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Women's Health and Education Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Bozkurt O, Uras N, Sari FN, Atay FY, Sahin S, Alkan AD, Canpolat FE, Oguz SS. Multi-dose vitamin d supplementation in stable very preterm infants: Prospective randomized trial response to three different vitamin D supplementation doses. Early Hum Dev. 2017 Sep;112:54-59. doi: 10.1016/j.earlhumdev.2017.07.016. Epub 2017 Aug 2. PMID 28779655